CLINICAL TRIAL: NCT02477748
Title: A 10-week Randomized, Multicenter, Double-blind, Parallel, Fixed-dose Study of MDX (Metadoxine Immediate-release/Slow-release, Bilayer Tablet) 1400 mg Compared With Placebo in Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: The MEASURE Study - A Phase 3 Study of MDX 1400 mg Daily Compared With Placebo in Adults With ADHD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: FDA Clinical hold
Sponsor: Alcobra Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL016
Record Dates: First submitted 2015-06-08; First posted 2015-06-23 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-04

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MDX (Active Comparator): Metadoxine Immediate-release/slow-release, bilayer tablet PO of 1400 mg, taken once daily for 10 weeks.; alternative name: MG01CI.
  Interventions: Drug: MDX
- Placebo (Placebo Comparator): Inert tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MDX — Immediate-release/slow-release,bilayer tablet PO of 1400 mg, taken once daily for 10 weeks.
  Other Names: MG01CI
  Arms: MDX
Drug: Placebo — Tablet PO, taken once daily for 10 weeks.
  Other Names: Inert tablet
  Arms: Placebo

SUMMARY:
This study is a multi-center, randomized, double-blind, placebo-controlled, phase 3 study of MDX (1400 mg daily) for 10 weeks compared with placebo in adults with ADHD.

The study will be comprised of Screening, Washout (if required), Treatment (total of 10 weeks) and Follow-up periods. Approximately 750 patients will be enrolled and undergo initial eligibility assessments.

DETAILED DESCRIPTION:
* A 10-week randomized, multi-center, double-blind, placebo-controlled, phase 3 study of MDX (1400 mg daily) for 10 weeks compared with placebo in adults with ADHD.
* The study will be comprised of Screening, Washout (if required), Treatment (total of 10 weeks) and Follow-up periods. Approximately 750 patients will be enrolled and undergo initial eligibility assessments.
* Subjects requiring a washout will undergo a Washout period where ADHD medication is discontinued (21 days for atomoxetine, 14 days for other ADHD medications). These subjects will have an Interim Visit (off drug) on or about Day -10 (Day -10 to Day -3) for CAARS-Inv assessment at the end of the Washout period.
* Subjects will be randomly assigned to placebo/MDX for a total treatment duration of up to ten weeks.

There will be a one week Follow-up period after the last dose of study treatment or early termination.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a man or a non-pregnant, non-lactating woman 18 to 55 years of age, inclusive, at the Screening visit.
2. Subject has a diagnosis of ADHD based on criteria in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM5) as assessed by the Adult ADHD Clinician Diagnostic Scale, (ACDS Version 1.2) modified for DSM-IV and DSM5 diagnoses; a diagnosis of ADHD not otherwise specified is unacceptable.
3. Male and Female subjects of childbearing potential must agree to use an effective contraceptive throughout the study
4. Subject is able to attend the clinic regularly and reliably.
5. Subject is able to swallow tablets and capsules.
6. Subject is able to understand, read, write, and speak the local language fluently to complete the study-related materials.
7. Subject is able to understand and sign an informed consent form to participate in the study.

Exclusion criteria

1. Subject has any current major psychiatric condition (e.g., schizophrenia, bipolar or personality disorder) or autism spectrum disorder.
2. Subject has any clinically significant or unstable medical or surgical condition that may preclude safe and complete study participation.
3. Subject has used an investigational medication/treatment or was enrolled in another clinical trial in the 30 days before the Screening visit.
4. Subject has used any medication or food supplement that the investigator or the medical monitor consider unacceptable during the 14-day period before the Baseline visit.
5. Subject's alcohol and caffeine intake will be assessed.
6. Subject has current suicidality, defined as active ideation, intent or plan, or any significant lifetime suicidal behavior (actual attempt, aborted attempt, interrupted attempt, or act or preparation towards imminently making a suicide attempt). Subjects exhibiting history (within previous 12 months) of non-suicidal self-injurious behavior will be excluded.
7. Subject has taken any prescription or non-prescription medication for ADHD during the 14 days (or 21 days for atomoxetine) before the Baseline visit. Subjects will not be allowed to take any other medications for ADHD besides the study medication (when prescribed) after the washout period and for the duration of the study, up to and including the safety Follow-up visit. (Other ADHD medications should NOT be prescribed to subjects before completion of the Follow-up visit or Early Termination Visit).
8. Subject is significantly visually impaired to an extent that is not able to be corrected by prescription glasses or contact lenses.
9. Subject is closely related to the sponsor, investigator, or study staff. Eligibility of subjects with any relationship to the sponsor, investigator, or study staff will be discussed with the medical monitor before study entry, and the medical monitor will decide on the eligibility of these cases.
10. Subject has previously been enrolled in an MDX clinical trial.
11. Subject lives in the same household as another subject in this clinical trial or in another on-going trial with MDX. Subject lives in the same household as someone who has previously participated in a trial with MDX.
12. Subject has any condition that, in the principal investigator's opinion, would place the subject at risk or influence the conduct of the study or interpretation of results, including (but not limited to) abnormally low intellectual capacity as judged by the investigator.
13. Subject cannot fully comprehend the implications of the protocol, cannot comply with its requirements, or is incapable of following the study schedule for any reason.
14. Subject is pregnant, lactating, or using an inadequate contraceptive method. Complete entry criteria will be reviewed and evaluated individually by a protocol trained delegate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 283 (Actual)
Dates: Start 2015-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
18-item total ADHD symptom score of the Conners Adult ADHD Rating Scale:O-SV (with the investigator as observer) with adult ADHD prompts (CAARS investigator). | 10 weeks
  The scale will be analyzed by change from Baseline to Week 10.

SECONDARY OUTCOMES:
Questionnaires of Clinical Global Severity of Illness (CGI-S) and Clinical Global Improvement (CGI-I). | 10 weeks
  The questionnaires will be analyzed by change from Baseline to all visits as well as by response rates.
Adult ADHD Self Report Scale (ASRS-Self) v1.1 Symptom Checklist - expanded version | 10 weeks
  The scale will be analyzed by change from Baseline to Week 10 in total score and sub- scales.
Test of Variables of Attention (TOVA) | 10 weeks
  A continuous performance test performed on the computer. Change from Baseline and response rate of Attention Comparison Score (ACS) will be assessed.
Test of Variables of Attention (TOVA) | 10 weeks
  A continuous performance test performed on the computer. Change from Baseline, as well as response rates, in variability of response time will be assessed.
Test of Variables of Attention (TOVA) | 10 weeks
  A continuous performance test performed on the computer. Change from Baseline, as well as response rates, in response time will be assessed.
Test of Variables of Attention (TOVA) | 10 weeks
  A continuous performance test performed on the computer. Change from Baseline, as well as response rates, in errors of commission will be assessed.
Test of Variables of Attention (TOVA) | 10 weeks
  A continuous performance test performed on the computer. Change from Baseline, as well as response rates, in errors of omission will be assessed.
Test of Variables of Attention (TOVA) | 10 weeks
  A continuous performance test performed on the computer. Change from Baseline, as well as response rates, in D-prime will be assessed.
Safety as assessed by adverse events (AEs) | 10 weeks
  Any undesirable experience associated with the use of a medical product in a subject
Safety as assessed by body temperature measurements | 10 weeks
  Body temperature measurements as part of vital signs measurements
Safety as assessed by Columbia Suicide Severity Rating Scale (C-SSRS) | 10 weeks
  C-SSRS scale allows investigators to gather lifetime history of suicidality as well as any recent suicidal ideation and/or behavior
Safety as assessed by laboratory tests; blood and urine | 10 weeks
  Laboratory test results (hematology, chemistry and urinalysis).
Safety as assessed by neurological evaluation | 10 weeks
  Neurological evaluation done by investigator
Safety as assessed by Electrocardiogram (ECG) test | 10 weeks
  Analysis and Interpretation of the Electrocardiogram
Safety as assessed by physical examinations | 10 weeks
  Physical examination done by investigator
Safety as assessed by discontinuations due to AEs | 10 weeks
  Discontinuations of subjects due to AEs
Safety as assessed by heart rate measurements | 10 weeks
  Heart rate measurements as part of vital signs measurements
Safety as assessed by respiratory rate measurements | 10 weeks
  Respiratory rate measurements as part of vital signs measurements
Safety as assessed by supine blood pressure | 10 weeks
  Supine blood pressure as part of vital signs measurements

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Newcorn, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (38):
- United States (36):
  - Harmonex, Inc., Dothan, Alabama
  - Pharmacology Research Institute, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, California
  - Artemis Institute for Clinical Research, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - MCB Clinical Research Centers, Colorado Springs, Colorado
  - Connecticut Clinical Research, Cromwell, Connecticut
  - Coastal Connecticut Research, New London, Connecticut
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Jacksonville, Florida
  - CNS Healthcare, Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - Institute for Advanced Medical Research, Alpharetta, Georgia
  - Goldpoint Clinical Research, Indianapolis, Indiana
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Rochester Center For Behavioral Medicine, Rochester Hills, Michigan
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - Premier Psychiatric Research Institute, Lincoln, Nebraska
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Global Medical Institutes, LLC, Princeton Medical Institute, Princeton, New Jersey
  - The Medical Research Network, New York, New York
  - Richard H Weisler, MD, PA, Raleigh, North Carolina
  - Neuro-Behavioral Clinical Research, Inc., Canton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Village Clinical Research Inc, Oklahoma City, Oklahoma
  - Summit Research Network, Portland, Oregon
  - Suburban Research Associates, Media, Pennsylvania
  - Carolina Clinical Research, Inc., Charleston, South Carolina
  - Clinical Neuroscience Solutions, Memphis, Tennessee
  - BioBehavioral Research of Austin at Specialty Clinic of Austin, Austin, Texas
  - Bayou City Research, Houston, Texas
  - Psychiatric & Behavioral Solutions, Salt Lake City, Utah
  - NeuroScience, Inc. (NSI), Herndon, Virginia
  - Summit Research Network(Seattle)LLC, Seattle, Washington
  - Dean Foundation - Middleton, Middleton, Wisconsin
- Israel (2):
  - Rambam Medical Center, Haifa
  - Geha Medical Centre, Petah Tikva

IPD SHARING:
Plan to Share IPD: No